CLINICAL TRIAL: NCT05563545
Title: A Phase Ⅰ Clinical Study on the Safety and Efficacy of Chimeric Antigen Receptor Gene Modified NK Cells Targeting CD19 in Patients With Recurrent or Refractory CD19 Positive Acute Lymphoblastic Leukemia
Brief Title: Anti-CD19 CAR-Engineered NK Cells in the Treatment of Relapsed/Refractory Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Simnova Biotechnology Co.,Ltd. (Industry)
Collaborators: Hebei Yanda Ludaopei Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XB-NK-1003
Record Dates: First submitted 2022-09-26; First posted 2022-10-03 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2022-09

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: NK; CD19 positive; Acute B lymphoblastic leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-NK-CD19 Cells (Experimental): After preconditioning with chemotherapy, CAR-NK-CD19 Cells will be evaluated.
  Interventions: Biological: CAR-NK-CD19 Cells

INTERVENTIONS:
Biological: CAR-NK-CD19 Cells — CAR-NK-CD19 Cells, 1-3×10^7 /KG, treatment follows a lymphodepletion. Drug: Fludarabine Recommendation: 25-30 mg/m2 (D-5~D-3), determined by tumor burden at baseline. Drug: Cyclophosphamide Recommendation: 250-300 mg/m2 (D-5~D-3), determined by tumor burden at baseline.

SUMMARY:
This study is a single arm clinical study to observe the safety ，dose tolerance and pharmacokinetic characteristics of CAR NK-CD19 in patients with recurrent or refractory CD19 positive acute lymphoblastic leukemia, and preliminarily evaluate the effectiveness, the immunogenicity of the product and the correlation between the changes of cytokines after infusion and CRS , ICANS.

DETAILED DESCRIPTION:
It is planned to select 9-21 patients with recurrent or refractory CD19 positive acute lymphoblastic leukemia （ALL）, from the lowest dose group. It is expected that 3-6 cases will be enrolled in each dose group. The protocol will be performed into screening period (-30~-10 days), prophase of lymophodepletion (-10~-5 days), Lymophodepletion (-5~-3 days), pre-infusion evaluation (-2~-1 days), infusion (day 0), and follow-up period (1-720 days). The incidence of DLT is observed after infusion. There are three preset dose groups in this clinical trial. The initial dose is 1.0 × 107 CAR positive NK cells/kg (body weight). Subsequent dose groups included 2.0 × 107 and 3.0 × 107 CAR positive NK cells/kg (body weight). The specific dose is determined by SRC based on the patient safety data and PK data. The maximum sample size of this study is tentatively 21 cases.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥12 years in the single-dose exploration phase, age ≥3 years in the dose exploration phase, both sexes;
* Meet the diagnostic criteria for recurrent or refractory CD19 positive acute lymphoblastic leukemia.
* The main organs have good organ function.
* The estimated survival time is ≥12 weeks.
* Blood pregnancy tests for women of childbearing age are negative.
* The patient himself/herself , and/or his/her legal guardian, agree to participate in the trial and sign the informed consent form.

Exclusion Criteria:

* Central nervous system involvement；
* Simple extramedullary leukemia or simple extramedullary recurrence；
* Received hematopoietic stem cell transplantation within the last 3 months and had graft-versus-host disease (GVHD) in the last 2 weeks, requiring immunosuppressive agents；
* Treated with high-dose corticosteroids in the last 1 week；
* Allogeneic cell therapy, major surgery, and live or attenuated vaccine had been received within 4 weeks prior to CAR NK-CD19 infusion；
* Had received other antitumor therapy or had an uncontrolled infection within 2 weeks prior to CAR NK-CD19 infusion；
* Systemic steroids were used within 3 days before CAR NK-CD19 infusion；
* Toxicity caused by previous treatment do not fully recover or do not stabilize to grade 1；
* Concomitant autoimmune diseases, central nervous system diseases, other active malignancies, infectious diseases, severe cardiovascular diseases, etc；
* Known allergies to study drugs or drugs that may be used in the study；
* Other conditions determined by Investigator which are not suitable for participation in the study

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2022-07-21 (Actual); Primary Completion 2022-11-25 (Actual); Study Completion 2022-11-25 (Actual)

PRIMARY OUTCOMES:
Safety of CAR NK-CD19 Cell | Up to 3 months after cell infusion
  Incidence of adverse events associated with CAR NK-CD19 treatment, abnormal clinically significant laboratory findings, including dose-limiting toxicity (DLT) and maximum-tolerated Dose (MTD).
Cell count of CAR NK-CD19 | From 1 to 720 days after infusion
  CAR NK-CD19 cell count
Cmax of CAR NK-CD19 | From 1 to 720 days after infusion
  CAR gene copy number maximum (Cmax)
Tmax of CAR NK-CD19 | From 1 to 720 days after infusion
  Time to maximum (Tmax)
AUC of CAR NK-CD19 | From 1 to 720 days after infusion
  Area under curve (AUC)
Other pharmacokinetic of CAR NK-CD19 Cell | From 1 to 720 days after infusion
  Other related pharmacokinetic parameters in peripheral blood and bone marrow

SECONDARY OUTCOMES:
The overall response rate (ORR) | Up to 3 months after cell infusion
  Total response rate (ORR) in 12 weeks (inclusive) after infusion of CAR NK-CD19 cells. CR/CRi ratio at 4 and 12 weeks; Duration of response (DOR); Progression free survival (PFS); Minimal residual disease (MRD) negative rate and duration at 4 and 12 weeks; Overall survival (OS)
Concentration of anti-drug antibody (ADA) | From 14 to 720 days after infusion
  Detection of anti-drug antibody (ADA) in CAR NK-CD19 cells
The changes of cytokines | Up to 3 months after cell infusion
  Detect the changes of cytokines in peripheral blood before and after CAR NK-CD19 cell infusion and the recovery time

CONTACTS AND LOCATIONS:
Locations (1):
- Hebei Yanda Ludaopei Hospital, Sanhe, Hebei, China